CLINICAL TRIAL: NCT01356745
Title: Efficacy of Premixed Nitrous Oxide and Oxygen in Patient With Out-of-hospital Moderate Acute Pain: a Randomized Double-blind Study
Brief Title: Efficacy of Premixed Nitrous Oxide and Oxygen in Patient With Out-of-hospital Moderate Acute Pain
Acronym: MEOPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0900603
Record Dates: First submitted 2010-06-22; First posted 2011-05-19 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Pain
Keywords: premixed nitrous oxide and oxygen; acute pain; prehospital setting
MeSH Terms: conditions — Acute Pain | interventions — Nitrous Oxide; Oxygen; kalinox; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- premixed 50% nitrous oxide and oxygen (Experimental)
  Interventions: Drug: Premixed 50% nitrous oxide and oxygen (Kalinox)
- medical air (Placebo Comparator)
  Interventions: Drug: medical air

INTERVENTIONS:
Drug: Premixed 50% nitrous oxide and oxygen (Kalinox) — 15 min inhalation dose (maximum duration of treatment of a subject)
  Arms: premixed 50% nitrous oxide and oxygen
Drug: medical air — inhalation gas for inhalation use
  Arms: medical air

SUMMARY:
Less than 10% of patients with a traumatic pain have been managed by a physician before to be admitted in an emergency service. 50 % of those patients have been carried by paramedics. Premixed nitrous oxide and oxygen is often used by paramedics, but no scientific studies have demonstrated its efficacy. The aim of the study is to demonstrate the efficacy of premixed nitrous oxide and oxygen in patients with out-of-hospital moderate acute pain.

DETAILED DESCRIPTION:
The study will evaluate the efficacy of premixed nitrous oxide and oxygen (MEOPA) in patients with out-of-hospital moderate acute pain.

The primary endpoint is the percentage of patients with pain relief (with a numerical rating scale of 3/10 or lower) 15 minutes after randomisation. Secondary endpoints are treatment safety and adverse events, time to analgesia and duration of analgesia. This study will expect 60 patients assigned in two parallel groups, defined by a randomization scheme. Group assignments were sealed in opaque envelopes and will be open sequentially by the dispatcher when the paramedic is ready to include the patient. The letter contained in the envelope corresponds to the cylinder to use. Eligible patients with a numeric rating scale (NRS) score between 3 and 6/10 are randomly allocated to receive either MEOPA, or medical air. Fifteen minutes after the randomisation, all patients will receive MEOPA from a distinct cylinder. Pain score will be measured at baseline and every 5 minutes until pain relief will be obtained. The paramedic blinded to the analgesic treatment groups will do all assessments of patients. The safety evaluation will include non invasive monitoring of blood pressure, heart rate, oxygen saturation by pulse oximetry (SpO2) and adverse events collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old
* Patients with a moderate acute pain (NRS score between 3 and 6)

Exclusion Criteria:

* Contraindication of premixed 50% nitrous oxide and oxygen
* Recent treatment of analgesic (less than 6 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with pain relief Number of patients with pain relief Number of patients with pain relief | 15 minutes
  Pain is mesured with a numerical rating scale (NRS)score on 10.Pain relief is defined by a NRS score of 3 or less

SECONDARY OUTCOMES:
Delay of analgesia (e.g. delay required to obtain analgesia) | Every 5 minutes from randomization for a one hour period
  Analgesia is obtained when the numerical rating scale score is or less than 3/10
Adverse events | Every 5 minutes from randomization for a one hour period
  Occurrence of any adverse event from a predefined list. Nausea, Emesis, Dizziness, Drowsiness, Dysphoria, Anxiety, Ear pain

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis DUCASSE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Universty Hospital Toulouse SAMU 31, Toulouse, France

REFERENCES:
- [Result] Ducasse JL, Siksik G, Durand-Bechu M, Couarraze S, Valle B, Lecoules N, Marco P, Lacombe T, Bounes V. Nitrous oxide for early analgesia in the emergency setting: a randomized, double-blind multicenter prehospital trial. Acad Emerg Med. 2013 Feb;20(2):178-84. doi: 10.1111/acem.12072. PMID 23406077